CLINICAL TRIAL: NCT06008093
Title: A Phase IIIb, Randomized, Multicenter, Open-label Study to Assess the Efficacy of Durvalumab Plus Tremelimumab Versus Pembrolizumab in Combination With Platinum-based Chemotherapy for First-line Treatment in Metastatic Non-small Cell Lung Cancer Patients With Non-squamous Histology Who Have Mutations and/or Co-mutations in STK11, KEAP1, or KRAS (TRITON)
Brief Title: A Study to Investigate the Efficacy of Durvalumab Plus Tremelimumab in Combination With Chemotherapy Compared With Pembrolizumab in Combination With Chemotherapy in Metastatic NSCLC Patients With Non-squamous Histology Who Have Mutations and/or Co-mutations in STK11, KEAP1, or KRAS
Acronym: TRITON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419ML00003
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Mutation; Metastatic Non-Small Cell Lung Cancer; Kelch-Like ECH-Associated Protein 1 (KEAP1); Kirsten rat sarcoma virus (KRAS); Programmed death-ligand 1 (PD-L1); Serine/threonine kinase 11 (STK11)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; tremelimumab; Pemetrexed; pembrolizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Phase IIIb 2-arm, parallel randomized open label multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Durvalumab + Tremelimumab + Platinum-based Chemotherapy (Experimental): Participants will receive durvalumab plus tremelimumab every 3 weeks (q3w) for four 21-day cycles in combination with chemotherapy followed by maintenance treatment period (durvalumab plus pemetrexed maintenance) every 4 weeks (q4w) until disease progression or unacceptable toxicity or treatment discontinuation. During the maintenance treatment period, participants will receive additional doses of tremelimumab at Cycle 6 (Week 16) and Cycle 28 (Week 104 - at Investigator's discretion) along with durvalumab and pemetrexed.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin
- Arm B: Pembrolizumab + Platinum-based Chemotherapy (Experimental): Participants will receive pembrolizumab regimen q3w for four 21-day cycles in combination with chemotherapy as induction treatment followed by maintenance treatment (pembrolizumab plus pemetrexed maintenance) q3w until disease progression or unacceptable toxicity or treatment discontinuation.
  Interventions: Drug: Pemetrexed; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Durvalumab — Participants will receive intravenous (IV) Durvalumab q3w for four 21-day cycles as induction treatment. Durvalumab will also be given during the maintenance treatment period q4w until disease progression or unacceptable toxicity.
  Other Names: MEDI4736 & IMFINZI®
  Arms: Arm A: Durvalumab + Tremelimumab + Platinum-based Chemotherapy
Drug: Tremelimumab — Participants will receive IV Tremelimumab q3w for four 21-days cycles as induction treatment. Tremelimumab will also be given during the maintenance therapy phase at week 16 and week 104 (at the investigators discretion).
  Other Names: IMJUDO®
  Arms: Arm A: Durvalumab + Tremelimumab + Platinum-based Chemotherapy
Drug: Pemetrexed — Participants in Arm A and Arm B will receive IV pemetrexed q3w for four 21-day cycles as induction treatment. In the maintenance therapy phase, Treatment Arm A will receive Pemetrexed q4w, Treatment Arm B will receive Pemetrexed q3w until disease progression or unacceptable toxicity.
  Other Names: Background Platinum-based Chemotherapy
Drug: Pembrolizumab — Participants will receive IV pembrolizumab q3w for four 21-days cycles as induction treatment. Pembrolizumab will also be given in the maintenance treatment phase q3w until disease progression or unacceptable toxicity or up to 24 months.
  Arms: Arm B: Pembrolizumab + Platinum-based Chemotherapy
Drug: Carboplatin — Participants will receive IV Carboplatin or IV Cisplatin on Day 1 of each 21-day cycle for 4 cycles as induction treatment.
  Other Names: Background Platinum-based Chemotherapy
Drug: Cisplatin — Participants will receive IV Carboplatin or IV Cisplatin on Day 1 of each 21-day cycle for 4 cycles as induction treatment.
  Other Names: Background Platinum-based Chemotherapy

SUMMARY:
The purpose of the study is to assess the efficacy of durvalumab plus tremelimumab in combination with chemotherapy compared with pembrolizumab in combination with chemotherapy in metastatic NSCLC patients with non-squamous histology who have mutations and/or co-mutations in STK11, KEAP1, or KRAS.

DETAILED DESCRIPTION:
A trial to learn if durvalumab plus tremelimumab with chemotherapy is safe and how well it works compared to pembrolizumab with chemotherapy in participants with metastatic non-small cell lung cancer with certain genetic mutations.

INFORMATION FOR TRIAL PARTICIPANTS:

Researchers are looking for a better way to treat people who have metastatic NSCLC and tumors with STK11, KEAP1, or KRAS genetic mutations. Most people learn they have NSCLC after it has already become metastatic, and it can no longer be treated with surgery.

Based on previous trials, researchers think durvalumab plus tremelimumab with chemotherapy could help participants more than the current standard treatment, which is pembrolizumab with chemotherapy. Durvalumab and tremelimumab are designed to work by helping the immune system recognize and kill cancer cells.

In this trial, researchers want to learn more about how well durvalumab plus tremelimumab with chemotherapy works in people with metastatic NSCLC and genetic mutations that can cause the cancer to be less responsive to treatment.

This trial is planned to have 280 participants. These participants will be randomly divided into one of two groups:

* One group will receive durvalumab plus tremelimumab with standard of care chemotherapy
* One group will receive pembrolizumab with standard of care chemotherapy

Durvalumab, tremelimumab, pembrolizumab, and chemotherapy are given as an injection over time into a vein, also called an IV infusion. Chemotherapy will be one of the following regimens: pemetrexed plus cisplatin or pemetrexed plus carboplatin.

This is an open-label trial. This means that each participant will know which trial treatment they receive, and the doctors and trial staff will also know.

Researchers will measure and compare:

* How long participants live during the trial
* How long participants live during the trial without their cancer getting worse
* How many participants' tumors respond to treatment
* How long participants' tumor responses last
* How long before participants need to start a different treatment type

Researchers will also keep track of all the medical problems participants have during the trial and monitor their safety.

Participants will stop receiving trial treatment if they no longer benefit from it or they stop participating for another reason.

Participants will visit their trial site every 3 to 4 weeks. At most visits, participants will:

* Have a physical exam and answer questions about any medications they are taking or any medical problems they have
* Receive their trial treatment
* Give blood and urine samples
* Have pictures of their tumors taken using CT or MRI scans

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented Stage IV non-squamous NSCLC not amenable to curative surgery or radiation.
* Participants must have tumors with STK11 or KEAP1 or KRAS mutations. Co-mutations are also allowed.
* Participants must have tumors that lack activating epidermal growth factor receptor mutations and ALK fusions.
* No prior chemotherapy or any other systemic therapy for metastatic NSCLC. Participants who have received prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation for advanced disease are eligible, provided that progression has occurred > 6 months from end of last therapy.
* No prior exposure to immune-mediated therapy excluding therapeutic anti-cancer vaccines, within 6 months of randomization.
* WHO/ECOG performance status of 0 or 1 at enrollment and randomization.
* Minimum life expectancy ≥ 12 weeks at randomization.
* At least 1 lesion, not previously irradiated, that qualifies as a RECIST 1.1 target lesion at baseline and can be accurately measured at baseline as ≥ 10 mm in the longest diameter with Computed Tomography (CT)/CT- Positron Emission Tomography or Magnetic Resonance Imaging and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines.
* Adequate organ and bone marrow function.
* Negative pregnancy test (urine or serum) for women of child-bearing potential
* Female participants must be 1 year post-menopausal, surgically sterile, or using one highly effective form of birth control
* Male and Female participants and their partners must use an acceptable method of contraception.
* Body weight of > 30 kg

Exclusion Criteria:

* Any evidence of acute or uncontrolled diseases or history of allogeneic organ transplant.
* Mixed small cell lung cancer and NSCLC histology.
* Major surgical procedure within 28 days prior to the first dose of the study intervention or an anticipated need for major surgery during the study.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], systemic lupus erythematosus, sarcoidosis, granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis [requiring immunosuppressive systemic therapy, eg, methotrexate, steroids], hypophysitis, uveitis, etc), autoimmune pneumonitis and autoimmune myocarditis. The following are exceptions to this criterion:

  * Participants with vitiligo or alopecia.
  * Participants with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Participants without active disease in the last 5 years may be included but only after consultation with the Study Clinical Lead.
  * Participants with celiac disease controlled by diet alone.
* Medical contraindication to platinum-based doublet chemotherapy.
* History of another primary malignancy except:

  * Malignancy treated with curative intent with no known active disease ≥ 2 years before the first dose of study intervention and of low potential risk for recurrence
  * Adequately resected non-melanoma skin cancer and curatively treated in situ disease.
* Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAE] Grade ≥ 2) caused by previous anti-cancer therapy, alopecia and vitiligo are excluded toxicities.
* Participants with Grade ≤ 2 neuropathy can be considered based on Investigator's judgement. Participants with irreversible toxicity that is not reasonably expected to be exacerbated by treatment with study intervention in the opinion of the Investigator may be included (eg, hearing loss).
* Spinal cord compression unless asymptomatic and stable.
* Participant meets the following:

  - Symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia (multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which requires treatment (CTCAE Grade 3), symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation controlled by medication or arrhythmias controlled by pacemakers may be permitted based on the Investigator judgement with cardiologist consultation recommended.
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (eg, hormone replacement therapy) is acceptable.
* No radiation therapy is allowed, unless it is 1) definitive radiation that had been administered at least 6 months prior, 2) palliative radiation to brain, with associated criteria for stability or lack of symptoms, or 3) palliative radiation to painful bony lesions (this must comprise less than 30% of the bone marrow)
* Patients with suspected brain metastases at screening should have an IV contrast-enhanced MRI (preferred) or IV contrast-enhanced CT/CT-PET of the brain prior to study entry. If brain metastases are detected patients must be treated before randomization. Randomization is only permitted if patients with brain metastases have:

  * Confirmed stable condition
  * Returned neurologically to baseline Brain metastases will not be recorded as RECIST target lesions at baseline.
* History of leptomeningeal carcinomatosis.
* Known to have tested positive for active tuberculosis infection
* Known active hepatitis infection, positive HCV antibody, HBsAg, or anti-HBc, at screening. Participants with a past or resolved HBV infection (defined as the presence of anti-HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if PCR is negative for HCV RNA. Participants co-infected with HBV and HCV, or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti-HBcAb with detectable HBV DNA); AND

  * HCV positive (presence of anti-HCV antibodies); OR
  * HDV positive (presence of anti-HDV antibodies).
* Known human immunodeficiency virus (HIV) infection that is not well controlled.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study intervention. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids or local steroid injections (eg, intra-articular injection).
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication, premedication for chemotherapy) or a single dose for palliative purpose (eg, pain control).
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
* Participants with a known hypersensitivity to any of the study interventions or any of the excipients of the products.
* For females only: Currently pregnant (confirmed with positive pregnancy test) or breastfeeding, or who are planning to become pregnant.

Female participants should refrain from breastfeeding from enrolment throughout the study and until up to 14 months after the last dose of cisplatin or 180 days after pemetrexed or 90 days after tremelimumab or durvalumab or pembrolizumab, whichever is longer; and during treatment with carboplatin.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-08-17 (Estimated); Study Completion 2031-03-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization until death, withdrawal of consent, or the end of the study (approximately 84 months)
  OS is defined as the time from randomization until death due to any cause in all participants. The measure of interest is the hazard ratio with corresponding 95% CI.
OS in subset of randomized participants with STK11 or KEAP1 mutations and/or co-mutations | From randomization until death, withdrawal of consent, or the end of the study (approximately 84 months)
  OS is defined as the time from randomization until death due to any cause in participants with STK11 or KEAP1 mutations and/or co-mutations. The measure of interest is the hazard ratio with corresponding 95% CI.

SECONDARY OUTCOMES:
Overall survival at 12 months | At 12 months
  OS is defined as the time from randomization until death due to any cause in all participants. The measure of interest is survival rate with corresponding 95% CI at 12 months landmark.
Overall survival at 24 months | At 24 months
  OS is defined as the time from randomization until death due to any cause in all participants. The measure of interest is survival rate with corresponding 95% CI at 24 months landmark.
Overall survival at 12 months in subset of randomized participants with STK11 or KEAP1 mutation and/or co mutations | At 12 months
  OS is defined as the time from randomization until death due to any cause. The measure of interest is survival rate with corresponding 95% CI at 12 months landmark.
Overall survival at 24 months in subset of randomized participants with STK11 or KEAP1 mutation and/or co mutations | At 24 months
  OS is defined as the time from randomization until death due to any cause. The measure of interest is survival rate with corresponding 95% CI at 24 months landmark.
Overall survival in subset of randomized participants whose PD-L1 status is PD-L1 TC < 1% | From randomization until death, withdrawal of consent, or the end of the study (approximately 84 months)
  OS is defined as the time from randomization until death due to any cause. The measure of interest is the hazard ratio with corresponding 95% CI.
Overall survival at 12 months in subset of randomized participants whose PD-L1 status is PD-L1 TC < 1% | At 12 months
  OS is defined as the time from randomization until death due to any cause. The measure of interest is survival rate with corresponding 95% CI at 12 months landmark.
Overall survival at 24 months in subset of randomized participants whose PD-L1 status is PD-L1 TC < 1% | At 24 months
  OS is defined as the time from randomization until death due to any cause. The measure of interest is survival rate with corresponding 95% CI at 24 months landmark.
Progression-free survival (PFS) | From randomization until disease progression, death, withdrawal of consent, or end of study (approximately 84 months)
  PFS is defined as the time from randomization until the date of confirmed PD (per Response Evaluation Criteria in Solid Tumours, Version 1.1 [RECIST 1.1] as assessed by the Investigator) or death due to any cause (in the absence of progression) in all participants. The measure of interest is the HR and the corresponding 95% CI.
Objective response rate (ORR) | From randomization until disease progression, or the last evaluable assessment in the absence of progression (approximately 84 months)
  ORR is defined as the proportion of participants with a confirmed objective tumour response (complete response [CR] or partial response [PR]) as determined by the investigator per RECIST 1.1 in all participants who have measurable disease at baseline. The measures of interest are the relative risk and common risk difference with corresponding 95% CI.
Duration of response (DOR) | From first documented response until documented progression (approximately 84 months)
  DOR is defined as the time from the date of first documented confirmed response until the date of documented progression (per RECIST 1.1, as assessed by the Investigator) or death due to any cause (in the absence of disease progression) in all participants who have confirmed objective response. The measure of interest is the median duration of response and corresponding 95% CI.
Time to First Subsequent Therapy (TFST) | From randomization until the start date of the first subsequent anti-cancer therapy after discontinuation of randomized study intervention or death [approx. up to 84 months]
  TFST is defined as the time from randomization until the start date of the first subsequent anti-cancer therapy after discontinuation of randomized study intervention, or death due to any cause in all participants. The measure of interest is the HR and the corresponding 95% CI.
Number of participants with adverse events (AEs) | From screening until the follow-up period is completed [approx. up to 84 months]
  To assess the safety and tolerability of durvalumab plus tremelimumab plus chemotherapy compared with pembrolizumab plus chemotherapy in participants with non-squamous histology who have metastatic NSCLC with mutations and/or co-mutations in STK11, KEAP1, or KRAS.

CONTACTS AND LOCATIONS:
Locations (85):
- United States (85):
  - Research Site, Birmingham, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Chandler, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Beverly Hills, California
  - Research Site, Irvine, California
  - Research Site, La Jolla, California
  - Research Site, Loma Linda, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Redding, California
  - Research Site, Santa Monica, California
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jupiter, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Albany, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Carterville, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Dyer, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Westwood, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Jamaica Plain, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Grand Island, Nebraska
  - Research Site, Lincoln, Nebraska
  - Research Site, Albany, New York
  - Research Site, Clifton Park, New York
  - Research Site, East Syracuse, New York
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Northport, New York
  - Research Site, Shirley, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Westbury, New York
  - Research Site, Bismarck, North Dakota
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Perrysburg, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Denton, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Kingwood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Skoulidis F, Borghaei H, Garon EB, Leal TA, Kaufman J, Liu SV, Nadler E, Patel SP, Peters S, Ricciuti B, Gautam A, Emeribe U, Luciani-Silverman L, Heymach JV. Rationale and design for a phase IIIb trial of first-line tremelimumab plus durvalumab versus pembrolizumab, in combination with chemotherapy, in patients with non-squamous metastatic non-small-cell lung cancer and mutations or co-mutations in STK11, KEAP1, or KRAS: the TRITON study. Ther Adv Med Oncol. 2025 Nov 6;17:17588359251386611. doi: 10.1177/17588359251386611. eCollection 2025. PMID 41209621